CLINICAL TRIAL: NCT04496219
Title: Acupuncture vs. Standard of Care for Induction Intravesical BCG-Related Adverse Events in High-Risk Non-Muscle Invasive Bladder Cancer
Brief Title: Acupuncture for the Treatment of Intravesical BCG-Related Adverse Events in High-Risk Non-muscle Invasive Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sarah Psutka, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1007421; P30CA015704 (NIH); NCI-2020-05021 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10544 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Bladder Urothelial Carcinoma In Situ; Recurrent Bladder Urothelial Carcinoma; Stage 0a Bladder Cancer AJCC v8; Stage 0is Bladder Cancer AJCC v8; Stage I Bladder Cancer AJCC v8; Superficial Bladder Urothelial Carcinoma
Keywords: Urinary Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Acupuncture Therapy; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (acupuncture, BCG) (Experimental): Patients undergo acupuncture therapy and receive BCG via intravesical injection on days 1, 8, 15, 22, 29, and 36 in the absence of unacceptable toxicity. Patients also receive standard of care symptom management.
  Interventions: Device: Acupuncture Therapy; Biological: BCG Solution; Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (BCG, standard of care) (Active Comparator): Patients receive BCG via intravesical injection on days 1, 8, 15, 22, 29, and 36 in the absence of unacceptable toxicity. Patients also receive standard of care symptom management. Patients may undergo acupuncture therapy after completion of intravesical BCG therapy.
  Interventions: Device: Acupuncture Therapy; Biological: BCG Solution; Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Device: Acupuncture Therapy — Undergo acupuncture therapy
  Other Names: Acupuncture
Biological: BCG Solution — Given by intravesical injection
  Other Names: Bacillus Calmette Guerin Solution; Bacillus Calmette-Guerin Solution; TICE BCG Solution
Other: Best Practice — Receive standard of care symptom management
  Other Names: standard of care; standard therapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the safety and feasibility of utilizing acupuncture in patients with high-risk bladder cancer that has not spread to the surrounding muscle (non-muscle invasive) undergoing treatment with Intravesical BCG. BCG is a weakened form of the bacterium Mycobacterium bovis that does not cause disease. It is used in a solution to stimulate the immune system in the treatment of bladder cancer. Unfortunately, many patients experience side effects such as pelvic pain, painful urination, severe urgency, frequency, urge incontinence, need to urinate at night, and/or infectious complications. These side effects may cause patients to delay or stop BCG treatment. Acupuncture is a medical intervention in which fine metallic needles are inserted into anatomical locations of the body to stimulate the peripheral and the central nervous system. Giving acupuncture before each intravesical BCG treatment may help to reduce the side effects of intravesical BCG, and help patients complete treatment. Specific outcomes of interest include acceptability to patients, effect of acupuncture on intravesical BCG-related side effects, and adverse events associated with acupuncture.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo acupuncture therapy and receive BCG via intravesical injection on days 1, 8, 15, 22, 29, and 36 in the absence of unacceptable toxicity. Patients also receive standard of care symptom management.

ARM II: Patients receive BCG via intravesical injection on days 1, 8, 15, 22, 29, and 36 in the absence of unacceptable toxicity. Patients also receive standard of care symptom management. Patients may undergo acupuncture therapy after completion of intravesical BCG therapy.

After completion of study, patients are followed up at 1 week.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Diagnosis of American Urological Association (AUA) high-risk non-muscle invasive bladder cancer (NMIBC), including high grade (HG) pT1 (invading only the lamina propria of the bladder), recurrent HG pTa (superficial tumors), HG pTa > 3 cm in size or multifocal, any carcinoma in situ, any variant histology, any lymphovascular invasion, and HG prostatic urethral involvement
* Diagnosis with urothelial carcinoma (primary histologic subtype), localized to the bladder, in the absence of nodal or other visceral metastases
* Patients who have been indicated for induction intravesical BCG in shared-decision-making with their primary urologist
* Have not received acupuncture in the previous 3 months
* Access to phone for study contacts
* Willing and able to participate in trial activities
* Platelets: 20,000/ uL or greater
* Absolute neutrophil count (ANC): 500 cells/uL or greater
* Able to understand and willing to sign written informed consent in English

Exclusion Criteria:

* Subjects who have had intravesical or systemic chemotherapy or radiation therapy for bladder cancer or for other malignancies prior to entering the study
* Subjects who are indicated to receive other intravesical agents or therapies concurrently with BCG will be excluded
* Subjects who have muscle-invasive bladder cancer, radiographic evidence of lymph node metastases or metastatic disease involving other organs including brain metastases
* Patients with predominant histology other than urothelial carcinoma of the bladder who would not otherwise be considered candidates for BCG
* BCG is contraindicated in:

  * Patients who are pregnant or lactating
  * Patients with active tuberculosis
  * Immunosuppressed patients with congenital or acquired immune deficiency, whether due to concurrent disease (e.g. acquired immunodeficiency syndrome [AIDS], lymphoma, leukemia), concomitant cancer therapy (cytotoxic drugs, radiation), or immunosuppressive therapy (e.g. corticosteroids, disease-modifying anti-rheumatic drugs [DMARDs])
  * Symptomatic urinary tract infection
  * Febrile illness
  * Patients requiring chronic treatment with certain antibiotics that may interfere with the effectiveness of BCG
  * Any previous allergies or severe reactions to BCG
* Not pregnant or trying to become pregnant. Acupuncture points included in the protocol are contraindicated with pregnancy
* Does not have a pacemaker. There is potential of electrostimulation interfering with the operation and function of pacemakers
* Patients requiring chronic treatment with certain antibiotics that may interfere with the effectiveness of BCG. Fluoroquinolone therapy may decrease the efficacy of intravesical BCG. Antibiotic therapy for ongoing treatment of active tuberculosis will decrease the efficacy of intravesical BCG
* Uncontrolled or concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded. Acupuncture points included in the protocol are contraindicated with pregnancy and BCG is contraindicated in pregnancy
* Pacemaker. Patients with pacemakers are restricted due to the potential of electrostimulation interfering with a pacemakers operation
* Platelets: < 20,000/ uL. Risk of bleeding with acupuncture
* ANC: < 500 cells/uL. Risk of infection with acupuncture
* Received acupuncture in the previous 3 months. Acupuncture treatment effects persist after a course of treatment, previous exposure to the intervention has the potential to affect the baseline data for treatment and control arms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah P. Psutka, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Acupuncture, BCG) | Arm II (BCG, Standard of Care)
Started | 28 | 17
Completed | 25 | 14
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Population: Some patients signed the consent but couldn't start the treatment because of progression of disease, those data were not collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Acupuncture, BCG) | Arm II (BCG, Standard of Care) | Total
Number analyzed (Participants) | 28 | 15 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 21 | 6 | 27
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72.6 [64.9 to 79] | 64.7 [59.6 to 75.3] | 70.27 [61.38 to 77.98]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 23 | 11 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 28 | 14 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 27 | 12 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 15 | 43
Smoking Status [Count of Participants; unit: Participants]
  Never | 8 | 1 | 9
  Former | 13 | 6 | 19
  Current | 1 | 6 | 7
  Unknown | 6 | 2 | 8
Tumor stage [Count of Participants; unit: Participants] — Pathologic stage Ta: Presence of a papillary tumor that does not infiltrate the bladder wall. Tis: The existence of carcinoma in situ, which constitutes a non-invasive flat high-grade (G3) cancer. T1: Tumor penetration into the connective tissue beneath the surface lining. All other stages were excluded. Ta is the least aggressive, and Tis and T1 are the most aggressive. Please note these were not outcomes, but were inclusion criteria for patients who would be eligible to receive induction BCG and therefore would be candidates for study entry.
  Participants
    pTis | 2 | 2 | 4
    pTa | 10 | 3 | 13
    pT1 | 15 | 6 | 21
    Unknown | 1 | 4 | 5
Charlson Comorbidity Index [Count of Participants; unit: Participants] — "The Charlson Comorbidity Index (CCI) was a method of categorizing comorbidities of patients based on the International Classification of Diseases diagnosis. The CCI score ranged from 0 (better outcome) to 21 (worse outcome). The higher the score, the more fragile/ill the patient was."
  Participants
    0 | 7 | 6 | 13
    1 | 5 | 3 | 8
    2 or greater | 16 | 6 | 22
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status criteria is used to assess how a patient's disease is progressing and to assess how the disease affects the daily living abilities of the patient. The scores on this instrument range from 0-5 (0=fully active and 5=dead), with higher scores indicating poorer performance.
  Participants
    0 | 7 | 9 | 16
    1 | 5 | 4 | 9
    2 | 16 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Trial Recruitment: Number of Participants Eligible, Enrolled, and Not Enrolled
Description: Will be described via qualitative report.
Time Frame: Up to 1 week after completion of treatment, an average of 7 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Screened for Trial Eligibility: Total number screened for trial eligibility
Arm/Group | Screened for Trial Eligibility
Number analyzed (Participants) | 50
Participants
  Eligible and agreed to participate | 45
  Did not meet inclusion criteria | 0
  Declined to participate | 3
  Regulatory hold 12/17/21-1/13/22 | 2

2. Primary Outcome: Trial Retention (Proportion Retained Versus All Enrolled, Reason for Not Completing)
Description: Will be described via qualitative report. Successful retention is defined as continued participation within the trial until 1 week following completion of induction.
Time Frame: Baseline, up to 1 week after completion of treatment, an average of 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Acupuncture, BCG) | Arm II (BCG, Standard of Care)
Number analyzed (Participants) | 28 | 17
Participants
  Number of enrolled and retained participants | 25 | 14
  Lost to follow-up: disease progression | 2 | 2
  Lost to follow-up: patient decision | 0 | 1
  Lost to follow-up: refractory hematuria | 1 | 0

3. Primary Outcome: Protocol Adherence (Proportion Adhered Versus All Enrolled, Specifics for How Protocol Was Not Followed and Why)
Description: Will be described via qualitative report. Protocol adherence is defined as completion of the acupuncture interventions and follow-up surveys if randomized to the acupuncture arm or completion of the follow-up surveys if randomized to the control arm.
Time Frame: Up to 1 week after completion of treatment, an average of 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Acupuncture, BCG) | Arm II (BCG, Standard of Care)
Number analyzed (Participants) | 28 | 17
Participants
  Protocol adherence | 17 | 8
  Missed visits due to UTI | 4 | 0
  Logistics/Scheduling Issues | 4 | 5
  Withdrew due to disease progression | 3 | 2
  Withdrew due to patient preference | 0 | 1
  Delay due to treatment of other comorbid condition | 0 | 1

4. Primary Outcome: Patient Satisfaction
Description: Patients' responses to the Cancer Care Satisfaction survey at 3 weeks and at the conclusion of induction Bacillus Calmette-Guerin (BCG) between two arms will be compared using t-test.
Time Frame: At 3 weeks and after completion of treatment, an average of 7 weeks
Population: Data were not collected
Arm/Group | Arm I (Acupuncture, BCG) | Arm II (BCG, Standard of Care)
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Clinic Staff's Responses to Surveys
Description: Clinic staff's responses to surveys assessing the healthcare burden of this protocol and time spent undergoing the acupuncture therapy for the experimental arm will be described via qualitative report
Time Frame: Up to 1 week after completion of treatment, an average of 7 weeks
Population: Data were not collected
Arm/Group | Arm I (Acupuncture, BCG) | Arm II (BCG, Standard of Care)
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Number of Adverse Events
Description: BCG related adverse events compared between patients receiving acupuncture and patients receiving standard of care.
Time Frame: Up to 1 week after completion of treatment, an average of 7 weeks
Population: The number of AEs are not mutually exclusive and participants may have reported more than one AE
Measure: Count of Units; unit: Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | Arm I (Acupuncture, BCG) | Arm II (BCG, Standard of Care)
Number analyzed (Participants) | 26 | 14
Number analyzed (Adverse Events) | 146 | 73
Adverse Events
  Bowel Symptoms | 14 | 5
  Fatigue | 36 | 15
  Flu-like Symptoms | 16 | 3
  Headache | 13 | 0
  Hematuria | 13 | 11
  Other | 8 | 4
  Pain | 9 | 11
  Urinary Symptoms | 37 | 24

7. Secondary Outcome: BCG Instillation Adherence (Out of a Possible Planned Six Treatments)
Description: BCG instillation adherence (successful adherence defined as the number of successfully administered BCG instillations of a possible 6 total) and weeks missed (measured as total weeks that BCG was not administered of the planned 6 weekly induction doses of intravesical BCG). Results between the acupuncture and control arms will be compared via t-test.
Time Frame: Up to 1 week after completion of treatment, an average of 7 weeks
Measure: Median (Inter-Quartile Range); unit: Visits
Arm/Group | Arm I (Acupuncture, BCG) | Arm II (BCG, Standard of Care)
Number analyzed (Participants) | 28 | 15
Visits
  Instillation adherence | 6 [6 to 7] | 6 [6 to 7]
  Missed visits | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); This p value relates to instillation adherence; Test type: Superiority; p = 0.97, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); This p value relates to missed visits; Test type: Superiority; p = 0.17, t-test, 2 sided

8. Secondary Outcome: Bladder and Bowel Symptoms as Self Reported by Patients
Description: Assessed using the EORTC - Non-Muscle Invasive Bladder Cancer 24 (EORTC-NMIBC24) symptom index, which was specifically designed to assess bladder and bowel symptoms for patients with NMIBC including assessments of impact of intravesical therapy. All of the subscales and single-item measures range in score from 0 to 100 and a high scale score represents a higher response level (ranging from 0 = low to 100 = high/healthy level of function; from 0 = low to 100 = high quality-of-life; from 0 = low to 100 = high level of symptomatology/problems). Subscale scores are each calculated by transforming individual item scores into a 0 to 1 scale, taking the mean, and multiplying by 100.
Time Frame: From week 1 to week 6 of treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm I (Acupuncture, BCG) | Arm II (BCG, Standard of Care)
Number analyzed (Participants) | 25 | 14
score on a scale
  Constipation Symptoms | 0 [0 to 0] | 0 [0 to 0]
  Diarrhea Symptoms | 0 [0 to 0] | 0 [-16.67 to 0]
  Urinary Symptoms | -9.52 [-21.43 to 0] | 0 [-8.33 to 9.52]
Statistical Analysis 1: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Constipation Symptoms; Test type: Superiority; p = 0.5638, Chi-squared
Statistical Analysis 2: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Diarrhea Symptoms; Test type: Superiority; p = 0.1753, Chi-squared
Statistical Analysis 3: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Urinary Symptoms; Test type: Superiority; p = 0.2062, Chi-squared

9. Secondary Outcome: Quality of Life: EORTC-QLQ-C30
Description: Assessed using the EORTC Health and Quality of Life Rating Scale (EORTC-QLQ-C30). All of the subscales and single-item measures range in score from 0 to 100 and a high scale score represents a higher response level (ranging from 0 = low to 100 = high/healthy level of function; from 0 = low to 100 = high quality-of-life; from 0 = low to 100 = high level of symptomatology/problems). Subscale and global health status scores are each calculated by transforming individual item scores into a 0 to 1 scale, taking the mean, and multiplying by 100.
Time Frame: From week 1 to week 6 of treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm I (Acupuncture, BCG) | Arm II (BCG, Standard of Care)
Number analyzed (Participants) | 25 | 14
score on a scale
  Global Health Organization | -8.33 [-16.67 to 0] | -4.17 [-16.67 to 0]
  Physical Function | 0 [-10 to 0] | 0 [-6.67 to 0]
  Emotional Function | 2.78 [0 to 16.67] | -4.17 [-12.5 to 12.5]
  Social Function | 0 [-16.67 to 0] | 0 [-16.67 to 0]
  Fatigue Symptoms | 0 [-11.11 to 0] | 0 [0 to 11.11]
  Pain Symptoms | 0 [-16.67 to 0] | 0 [-16.67 to 0]
  Malaise Symptoms | 0 [-16.67 to 0] | 0 [0 to 8.33]
  Role Function | 0 [0 to 0] | 0 [-16.67 to 0]
  Cognitive Function | 0 [-16.67 to 0] | 0 [-16.67 to 8.33]
  Nausea Symptoms | 0 [0 to 0] | 0 [0 to 0]
  Dyspnoea Symptoms | 0 [0 to 0] | 0 [0 to 0]
  Insomnia Symptoms | 0 [-33.33 to 33.33] | 0 [-16.67 to 0]
  Appetite Loss Symptoms | 0 [0 to 0] | 0 [0 to 0]
  Finances | 0 [0 to 0] | 0 [0 to 0]
  Intravesical Symptoms | 0 [0 to 0] | 0 [0 to 0]
  Worries | -11.11 [-20.83 to 0] | -8.33 [-16.67 to 0]
  Bloating Symptoms | 0 [-16.67 to 0] | -8.33 [-16.67 to 0]
  Sexual Function | 0 [-16.67 to 0] | 0 [0 to 16.67]
  Male Sex Problems | 0 [-16.67 to 0] | 0 [-16.67 to 0]
  Intimacy | 0 [-33.33 to 0] | 0 [-33.33 to 0]
Statistical Analysis 1: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Global Health; Test type: Superiority; p = 0.8092, Chi-squared
Statistical Analysis 2: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Physical Function; Test type: Superiority; p = 0.5492, Chi-squared
Statistical Analysis 3: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Emotional Function; Test type: Superiority; p = 0.6464, Chi-squared
Statistical Analysis 4: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Social Function; Test type: Superiority; p = 0.586, Chi-squared
Statistical Analysis 5: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Fatigue Symptoms; Test type: Superiority; p = 0.8999, Chi-squared
Statistical Analysis 6: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Pain Symptoms; Test type: Superiority; p = 0.2007, Chi-squared
Statistical Analysis 7: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Malaise Symptoms; Test type: Superiority; p = 0.9921, Chi-squared
Statistical Analysis 8: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Role Function; Test type: Superiority; p = 0.5723, Chi-squared
Statistical Analysis 9: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Cognitive Function; Test type: Superiority; p = 0.812, Chi-squared
Statistical Analysis 10: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Nausea Symptoms; Test type: Superiority; p = 0.96, Chi-squared
Statistical Analysis 11: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Dyspnoea Symptoms; Test type: Superiority; p = 0.1062, Chi-squared
Statistical Analysis 12: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Insomnia Symptoms; Test type: Superiority; p = 0.3259, Chi-squared
Statistical Analysis 13: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Appetite Loss Symptoms; Test type: Superiority; p = 0.9664, Chi-squared
Statistical Analysis 14: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Finances; Test type: Superiority; p = 0.4564, Chi-squared
Statistical Analysis 15: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Intravesical Symptoms; Test type: Superiority; p = 0.1036, Chi-squared
Statistical Analysis 16: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Worries; Test type: Superiority; p = 0.1789, Chi-squared
Statistical Analysis 17: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Bloating Symptoms; Test type: Superiority; p = 0.5186, Chi-squared
Statistical Analysis 18: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Sexual Function; Test type: Superiority; p = 0.0757, Chi-squared
Statistical Analysis 19: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Male Sex Problems; Test type: Superiority; p = 0.1174, Chi-squared
Statistical Analysis 20: Comparison: Arm I (Acupuncture, BCG) vs Arm II (BCG, Standard of Care); For the patient survey, the two arms will be compared using chi-squared. This analysis is for Intimacy; Test type: Superiority; p = 0.3129, Chi-squared

10. Secondary Outcome: Median Weekly Pill Counts of Medications Prescribed for the Management of BCG-related Side Effects, Standardized by Dosage Across Medication Types
Description: Will be compared via Wilcoxon rank sum test.
Time Frame: Up to 1 week after completion of treatment, an average of 7 weeks
Population: Data were not collected
Arm/Group | Arm I (Acupuncture, BCG) | Arm II (BCG, Standard of Care)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of first exposure to acupuncture through the end of treatment, an average of 7 weeks, on a weekly basis. BCG related adverse events were compared between patients receiving acupuncture and patients receiving standard of care and were recorded up to 1 week after completion of treatment, an average of 7 weeks.
Description: Toxicity or AEs related to BCG administration were collected by patient survey on a weekly basis using the CTCAE v.50 assessment of Systemic Therapy Toxicity. Patients in the acupuncture arm were surveyed weekly prior to acupuncture treatments regarding side effects and potential adverse events associated with the acupuncture intervention using the CTCAE v5. There were two acupuncture-related adverse events: 1 patient reporting a Grade 1 bruise and 1 patient reporting a Grade 1 pain.
Arm/Group | Arm I (Acupuncture, BCG) | Arm II (BCG, Standard of Care)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/14
Other Adverse Events (participants affected / at risk) | 24/26 | 14/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Acupuncture, BCG) (N=26) | Arm II (BCG, Standard of Care) (N=14)
Bruise (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bowel Symptoms (Gastrointestinal disorders) | 9 (14) | 3 (5)
Fatigue (General disorders) | 15 (36) | 6 (15)
Flu-like Symptoms (General disorders) | 9 (16) | 3 (3)
Headache (Nervous system disorders) | 10 (13) | 0 (0)
Hematuria (Renal and urinary disorders) | 9 (13) | 6 (11)
Pain (Musculoskeletal and connective tissue disorders) | 7 (10) | 6 (11)
Urinary Symptoms (Renal and urinary disorders) | 16 (37) | 11 (24)
Other (General disorders) | 8 (8) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT04496219/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT04496219/ICF_000.pdf